CLINICAL TRIAL: NCT07373496
Title: Pilot Study of a Novel Patient Position Monitoring System for Beam Gated Radiation Therapy of Malignancies of the Chest and Upper Abdomen
Brief Title: Patient Position Monitoring System for Beam Gated Radiation Therapy of Malignancies of the Chest and Upper Abdomen
Status: Not yet recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: EmpNia (Unknown)
Responsible Party: Sponsor
Other Study IDs: 202512129
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Radiotherapy; Radiotherapy, Image-Guided
Keywords: Radiotherapy; Cancer; Motion
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Motion management system during standard of care treatment: Patients will wear the motion management system (eMotus) during their CT simulation scan and each of their radiation therapy treatments (no more than 15 fractions). CT simulation will take approximately 40 minutes and radiation treatments will take approximately 15-45 minutes depending on the patient's plan. Patients will complete questionnaires collecting feedback on the device after receiving their last fraction of treatment.
  Interventions: Device: Patient Position Monitoring System

INTERVENTIONS:
Device: Patient Position Monitoring System — The device is a motion management system for patients receiving radiation therapy. The system is composed of a disposable fiber optic sensor pad, a signal transceiver, and software to receive and display patient data. The sensor pad is applied to the patient's chest or abdomen and plugged into the signal transceiver, which provides the system's software to provide a visual respiratory trace for the treatment team.
  Other Names: EmpNia eMotus

SUMMARY:
This study will evaluate the feasibility of using this novel patient position monitoring system for patients receiving radiation therapy to targets involving the chest or upper abdomen, as these are the most affected by respiratory motion. This motion monitoring system will be incorporated with standard of care on-board CT imaging to confirm that the respiratory position is tracking the tumor target appropriately.

ELIGIBILITY:
Eligibility Criteria

* Planning to receive a course of radiation therapy that, per the treating radiation oncologist, requires motion management at the time of CT simulation and during treatment. Types of treatments that require motion management during radiation therapy include treatments to the lung, heart, breast, and upper abdomen (pancreas, liver, adrenals). These may include either free-breathing treatments or breath-hold treatments.
* At least 18 years of age.
* No documented allergy to medical grade adhesives.
* Able to understand and willing to sign an IRB approved written informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who will be receiving standard of care radiation therapy approaches for tumors involving the chest wall (ribs, soft tissue, breast), thorax (lung, heart), or upper abdomen (liver, adrenal glands, pancreas, para-aortic lymph nodes) that requires motion management at Washington University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Feasibility of eMotus system as defined by frequency of successfully delivered treatment fraction | Enrollment to completion of radiation therapy (estimated total time is 1 month)
  The feasibility of the eMotus fiber optic motion sensor system will be measured as the frequency of scheduled treatment fractions delivered successfully using eMotus. Success is defined as delivery of a treatment fraction in one on-table attempt without requiring the use of a secondary (backup) motion management system. Unsuccessful delivery of a treatment fraction will be defined as more than one attempt for gating without reproducible positioning, breath-hold, or surface guidance feedback such that the treatment could not be delivered with eMotus. Descriptive statistics will be collected and reported to determine the proportion of successful motion monitoring events.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Samson, MD, MPHS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal can email the Principal Investigator at psamson@wustl.edu. To go access, data requestors will need to sign a data access agreement.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu